CLINICAL TRIAL: NCT03164499
Title: Effectiveness of an Intensive Intervention to Improve Lifestyles in Subjects With Intermediate Cardiovascular Risk: a Randomized Controlled Trial.
Brief Title: Intensive Intervention to Improve Lifestyles in Subjects With Intermediate Cardiovascular Risk.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BIO 16/00006
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Risk Factor
Keywords: Health education; Life style; Risk factors; Cardiovascular diseases; Cognitive performance; Quality of life
MeSH Terms: conditions — Health Education; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Individual counselling on lifestyles.
  Interventions: Behavioral: Individual counselling on lifestyles
- Intervention group (Experimental): Individual counselling on lifestyles and additional group counselling on lifestyles.
  Interventions: Behavioral: Individual counselling on lifestyles; Behavioral: Additional group counselling on lifestyles

INTERVENTIONS:
Behavioral: Individual counselling on lifestyles — Individual standardized counselling on healthy diet, daily physical activity, stress management, smoking cessation, and moderation in alcohol consumption.
Behavioral: Additional group counselling on lifestyles — Group sessions focusing on cardiovascular risk, diet and moderation in alcohol consumption, physical activity and stress management, and smoking cessation will be held in health centres for four consecutive weeks. Each session will last 60-90 minutes, and will be led by two trained nurse practitioners. Ten participants will assist each group. During each session, attendance will be recorded and printed educational materials related to the topic addressed will be distributed.
  Follow-up calls to reinforce lifestyle modification and record the barriers to behaviour change found will be performed 6 and 9 months after enrolment.
  Arms: Intervention group

SUMMARY:
This is a randomized controlled trial aimed to design an intensive intervention to modify lifestyles of subjects with intermediate cardiovascular risk and evaluate its effectiveness. 200 participants aged 35-74 years who have intermediate cardiovascular risk will be included. Subjects will be selected by consecutive sampling at urban primary care health centers from Salamanca (Spain) and they will be randomized to a control or an intervention group. Both groups will receive individual standardized counselling on healthy diet, daily physical activity, smoking cessation, and moderation in alcohol consumption. Moreover, individuals from the intervention group will receive additional group counselling and follow-up calls. The effect of the intervention will be assessed using lifestyles and quality of life questionnaires, metabolic control parameters, inflammation markers, anthropometric and vascular function measurements, and neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 35-74 years who had an intermediate cardiovascular risk defined according to the Framingham risk equation will be included.

Exclusion Criteria:

* Personal history of atherosclerotic disease.
* Unable to do exercise or follow the Mediterranean diet.
* Institutionalized.
* Terminal illness.
* Mental disorders that limited the intervention compliance.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Adherence to the Mediterranean diet | 1 year
  Measurement by validated 14-point Mediterranean Diet Adherence Screener
Self-reported physical activity | 1 year
  Measurement by short version of the International Physical Activity Questionnaire

SECONDARY OUTCOMES:
Changes in physical activity | 1 year
  Measurement by Pedometer
Changes in dietary pattern | 1 year
  Measurement by semi-quantitative Food Frequency Questionnaire
Cardiovascular risk factors | 1 year
  Measurement by Framingham Risk Score
Body composition | 1 year
  Measurement by Bioelectrical Impedance Analyzer
Cardio-ankle vascular index (CAVI) | 1 year
  Measurement by Vasera® VS-2000 device
Brachial-ankle pulse wave velocity (ba-PWV) | 1 year
  Measurement by Vasera® VS-2000 device
Ankle-brachial index (ABI) | 1 year
  Measurement by Vasera® VS-2000 device
Health related quality of life | 1 year
  Measurement by Spanish version of the SF-12 questionnaire
Immediate verbal memory | 1 year
  Assessment by immediate recall of a list of 15 words, in three attempts
Delayed verbal memory | 1 year
  Assessment by free recall of the words learnt in the first part of the study after a period of approximately 10 minutes
Phonological fluency | 1 year
  Assessment by enumerating for one minute as many words as possible starting with different letters
Attention | 1 year
  Assessment by Trail Making Test A
Processing speed | 1 year
  Assessment by Trail Making Test B
Executive functions | 1 year
  Assessment by Trail Making Test B
Working memory | 1 year
  Assessment by WAIS Digit Span Backward test
Sustained attention | 1 year
  Assessment by Stroop test
Selective attention | 1 year
  Assessment by Stroop test

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mora Simón, PhD, Principal Investigator — Primary Care Research Unit, The Alamedilla Health Center
Locations (1):
- Primary Care Research Unit, The Alamedilla Health Center, Salamanca, Castilla and Leon, Spain